CLINICAL TRIAL: NCT00329485
Title: The Effect of Ribose on B-Type Natriuretic Peptide Levels in Congestive Heart Failure Patients
Brief Title: The Effect of Ribose on B-Type Natriuretic Peptide (BNP) Levels in Congestive Heart Failure Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Poor recruitment and through put
Sponsor: Valen Labs (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: 200602-WA; WIRB Study No. 1076926
Record Dates: First submitted 2006-05-23; First posted 2006-05-24 (Estimated); Last update posted 2007-08-02 (Estimated); Status verified 2007-08

CONDITIONS: Congestive Heart Failure
Keywords: Elevated BNP Levels in CHF patients
MeSH Terms: conditions — Heart Failure | interventions — Ribose

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: CORvalen (D-Ribose)

SUMMARY:
The purpose of this research study is to test the effectiveness of CORvalen, a medical food, to increase cellular energy sufficiently to change or modify BNP levels in congestive heart failure patients.

DETAILED DESCRIPTION:
B-type natriuretic peptide (BNP), is a blood test commonly used to track the progress of congestive heart failure. CORvalen, a medical food, contains D-Ribose (ribose), a natural substance that has been shown to improve the amount of energy compounds at the cellular level. Congestive heart failure has been associated with a reduced level of high-energy compounds. One researcher has called them an "energy starvation" in congestive heart failure. This study will try to assess if increasing the amount of these energy compounds is sufficient to improve BNP levels. Approximately 120 symptomatic congestive heart failure patients will participate in this 3 month study.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic adults, M/F, between 18 and 80 years of age
* BNP levels equal to or greater than 300 pg/ml.
* Primary or secondary diagnosis of congestive heart failure at the time of admission (any NYHA Class)
* Diagnosis of congestive heart failure for at least 3 months
* Able to perform 6 minute hall walk
* No therapeutic pharmaceutical class changes for at least 1 month
* Provide informed consent
* A 30-day washout period must be achieved for any patient involved in a previous clinical study.

Exclusion

* Insulin dependent diabetes (Type I)
* History of obstructive valvular disease
* History of pulmonary hypertension within the last 3 months
* History of hypertrophic or alcoholic cardiomyopathy
* History of restrictive cardiomyopathy
* History of reversible cardiomyopathy
* History of non-compliance
* Pregnancy
* Current enrollment in any other clinical study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120
Dates: Start 2006-06; Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Demonstrate a significant reduction in serial BNP values over 3 months while on ribose supplementation

SECONDARY OUTCOMES:
Demonstrate significant improvement in serial six minute hall walks while on ribose supplementation
Demonstrate significant improvement in quality of life as measured by the Minnesota, Living with Heart Failure Questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Garrie Haas, MD, Principal Investigator — Ohio State University; Mark Munger, PharmD, Principal Investigator — University of Utah; Reynolds Delgado, MD, Principal Investigator — Texas Heart Institute; Daniel Pauly, MD, PhD, Principal Investigator — University of Florida; Kris Vijay, MD, Principal Investigator — Scottsdale Cardiovascular Research Institute; Masoor Kamalesh, MD, Principal Investigator — Roudebush VA Medical Center; Robert J Weiss, MD, Principal Investigator — Maine Research Associates
Locations (1):
- See list of Study Principal Investigators, Columbus, Ohio, United States